CLINICAL TRIAL: NCT01590641
Title: A Double-Blind, Randomized, Placebo-Controlled, Single and Multiple- Dose Ranging, Adaptive Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Antiviral Activity of GS-9620 in Treatment Naive Subjects With Chronic Hepatitis B Virus Infection
Brief Title: A Study Evaluating GS-9620 in Treatment Naive Subjects With Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-283-0106
Record Dates: First submitted 2012-04-30; First posted 2012-05-03 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Hepatitis B; HBV
Keywords: Hepatitis; Hepatitis B; Hepatitis B Virus; HBV; GS-9620; Toll-like receptor (TLR)-7 Agonist
MeSH Terms: conditions — Hepatitis B; Hepatitis | interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide; Cohort Studies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 0.3mg GS-9620 (Experimental)
  Interventions: Drug: Single Ascending Dose (SAD) Cohorts GS-9620
- 1mg GS-9620 (Experimental)
  Interventions: Drug: Single Ascending Dose (SAD) Cohorts GS-9620
- 2mg GS-9620 (Experimental)
  Interventions: Drug: Single Ascending Dose (SAD) Cohorts GS-9620
- 4mg GS-9620 (Experimental)
  Interventions: Drug: Single Ascending Dose (SAD) Cohorts GS-9620
- 0.3mg GS-9620 QW x 2 doses (Experimental)
  Interventions: Drug: Multiple Ascending Dose (MAD) Cohorts
- 1mg GS-9620 QW x 2 doses (Experimental)
  Interventions: Drug: Multiple Ascending Dose (MAD) Cohorts
- 2mg GS-9620 QW x 2 doses (Experimental)
  Interventions: Drug: Multiple Ascending Dose (MAD) Cohorts
- 4mg GS-9620 QW x 2 doses (Experimental)
  Interventions: Drug: Multiple Ascending Dose (MAD) Cohorts

INTERVENTIONS:
Drug: Single Ascending Dose (SAD) Cohorts GS-9620 — This study will enroll cohorts of 6 eligible, unique subjects per cohort, randomized to either active drug or placebo (5:1) within each cohort. Subjects in Single Ascending Dose (SAD) Cohorts will receive a single dose of GS-9620.
  Arms: 0.3mg GS-9620; 1mg GS-9620; 2mg GS-9620; 4mg GS-9620
Drug: Multiple Ascending Dose (MAD) Cohorts — This study will enroll cohorts of 6 eligible, unique subjects per cohort, randomized to either active drug or placebo (5:1) within each cohort. Subjects in Multiple Ascending Dose (MAD) Cohorts will receive GS-9620 once weekly for two weeks (QW x 2 doses)
  Arms: 0.3mg GS-9620 QW x 2 doses; 1mg GS-9620 QW x 2 doses; 2mg GS-9620 QW x 2 doses; 4mg GS-9620 QW x 2 doses

SUMMARY:
Dose cohorts may be dosed with one of up to 4 possible total weekly doses (0.3 mg, 1 mg, 2 mg, 4 mg). Dose escalation or repetition will be governed by pre-specified safety and activity rules. Subjects will be confined on either days 1-3 or days 1-3 and 8-10. Follow-up visits are also required periodically through day 43, and potential viral load follow-up visits at weeks 3 and 6 months post last dose. Study procedures involve blood draws for pharmacokinetic, pharmacodynamic, virologic, and safety assessments

ELIGIBILITY:
Inclusion Criteria:

* Chronic HBV infection ≥ 6 months
* HBsAg ≥ 250 IU/mL
* HBV treatment naïve
* Absence of extensive bridging fibrosis (Metavir 3 or greater) or cirrhosis
* Creatinine clearance ≥ 70 mL/min

Exclusion Criteria:

* Co-infection with hepatitis C virus (HCV), hepatitis D virus (HDV), or HIV
* History of Gilberts disease
* Laboratory parameters not within defined thresholds for leukopenia, neutropenia, anemia, thrombocytopenia, thyroid-stimulating hormone (TSH), or other evidence of hepatic decompensation
* Diagnosis of autoimmune disease, poorly controlled diabetes mellitus, significant psychiatric illness, severe chronic obstructive pulmonary disease(COPD), malignancy, hemoglobinopathy, retinal disease, or patients who are immunosuppressed
* Evidence of hepatocellular carcinoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events in single and multiple oral doses of GS-9620 | Periodically Through Week 25
  Safety will be assessed during the study through the reporting of adverse events, by clinical laboratory tests, physical examinations including vital signs and ECGs at various time points during the study, and by documentation of concomitant medications throughout the study.

SECONDARY OUTCOMES:
Assessment of plasma drug concentrations of GS-9620 using non-compartmental methods | Day 1 and Day 8
  Single ascending dose (SAD) and multiple ascending dose (MAD) Cohorts:serial blood samples will be collected on Day 1 at 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48, and 96 hours post-dose.
  MAD Cohorts: serial blood samples will also be collected on Day 8 at 0 (pre-dose), , 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hours post-dose.
Measurement of pharmacodynamic markers (cytokines and interferon-stimulated genes [ISGs]) | Up to Day 15
  SAD Cohorts: whole blood and serum for pharmacodynamic (PD) assessments (RNA and cytokine analysis) will be drawn on Day 1: pre-dose and 8-hr post dose, Day 2, Day 3, Days 5 and Day 8
  MAD Cohorts: whole blood and serum for PD assessments (RNA and cytokine analysis) will be drawn on Day 1: pre-dose and 8 hours postdose, Day 2, Day 3, Day 5, and Day 8: pre-dose and 8 hours post-dose, Day 9, Day 10, Day 12, and Day 15
Reduction of hepatitis B (HBV) viral load from baseline | Up to Day 15 and Follow-Up
  Antiviral activity will be evaluated by determination of HBV HBsAg and HBV viral load kinetics

CONTACTS AND LOCATIONS:
Overall Officials: Benedetta Massetto, M.D., Study Director — Gilead Sciences
Locations (23):
- United States (13):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - West Coast Clinical Trials, LLC, Costa Mesa, California
  - University of California Antiviral Research Center (AVRC), San Diego, California
  - Indiana University Medical Center, Indianapolis, Indiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - Weill Cornell Medical College, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Australia (4):
  - Nepean Hospital, Kingswood, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Monash University, Department of Medicine, Clayton, Victoria
  - Royal Perth Hospital, Nedlands, Western Australia
- Canada (3):
  - University of Calgary, Heritage Medical Research Center, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Algorithme Pharma, Inc., Montreal, Quebec
- Auckland Clinical Studies, Grafton, Auckland, New Zealand
- South Korea (2):
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul